CLINICAL TRIAL: NCT01328938
Title: A Randomized,Multi-center,Parallel-group, Phase II(Single-blind)/Phase III(Double- Blind)Study to Determine the Optimal Dose and to Evaluate the Efficacy and Safety of GCPGC on Chemotherapy-induced Neutropenia Compared to Neulasta(Pegfilgrastim)
Brief Title: GCPGC in Chemotherapy-induced Neutropenia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Green Cross Corporation (Industry)
Collaborators: Symyoo (Industry)
Responsible Party: Sponsor
Organization: GC Biopharma Corp (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: GCPGC P2/3
Record Dates: First submitted 2011-02-06; First posted 2011-04-05 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2013-11

CONDITIONS: Chemotherapy Induced Neutropenia
Keywords: Pegfilgrastim; neutropenia
MeSH Terms: conditions — Neutropenia | interventions — pegfilgrastim

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Stage I - Arm I: GCPGC I (3.6mg) (Experimental): GCPGC 3.6mg, sc, once at Day 2 per cycle (in patients receiving chemotherapy at Day 1)
  Interventions: Biological: GCPGC 3.6mg
- Stage I - Arm II: GCPGC II (6mg) (Experimental): GCPGC 6mg, sc, once at Day 2 per cycle (in patients receiving chemotherapy at Day 1)
  Interventions: Biological: GCPGC 6mg
- Stage II - Arm I: GCPGC (Experimental): GCPGC 6mg, sc, once at Day 2 per cycle (in patients receiving chemotherapy at Day 1).
  The recommended dose in Stage II was determinated as GCPGC 6mg in Stage I.
  Interventions: Biological: GCPGC 6mg
- Stage II - Arm II: Neulasta (Active Comparator): Neulasta 6mg, sc, once at Day 3 per cycle (in patients receiving chemotherapy at Day 1)
  Interventions: Biological: Neulasta (pegfilgrastim) 6mg

INTERVENTIONS:
Biological: GCPGC 3.6mg — Stage I:Single blinded
  Other Names: Pegfilgrastim
  Arms: Stage I - Arm I: GCPGC I (3.6mg)
Biological: GCPGC 6mg — Stage I: Single blinded;
  Other Names: Pegfilgrastim
  Arms: Stage I - Arm II: GCPGC II (6mg)
Biological: Neulasta (pegfilgrastim) 6mg — Stage II: Active comparator, double blinded
  Arms: Stage II - Arm II: Neulasta
Biological: GCPGC 6mg — Experimental: Stage II
  Other Names: Pegfilgrastim
  Arms: Stage II - Arm I: GCPGC

SUMMARY:
This study is adaptive design and it consists of stage I and stage II.

Stage I is multi-center, parallel-group, single-blind, phase II study to determine the adequate dose of GCPGC in chemotherapy-induced neutropenia. 2 Different doses of GCPGC will be investigated in a total of 60 Breast cancer patients who are receiving chemotherapy.

Stage II is multi-center, parallel-group, double-blind,phase III study to evaluate the efficacy and safety of once per cycle GCPGC in chemotherapy-induced neutropenia compared to Neulasta (pegfilgrastim). A total of 120 patients receiving chemotherapy will participate into this phase.

DETAILED DESCRIPTION:
GCPGC ia a solution for containing pegfilgrastim. Pegfilgrastim is a covalent conjugate of recombinant human granulocyte colony-stimulating factor (G-CSF) with a polyethylene glycol (PEG) which has long half life compared to filgrastim, resulting in dosing advantage.

ELIGIBILITY:
Inclusion Criteria:

* women(≥ 18 years old) diagnosed with breast cancer who are receiving chemotherapy inducing neutropenia
* body weight of 45kg and more
* ECOG performance status 2 and less
* ANC ≥1,500mm3 and Platelet ≥100,000/mm3
* life expectancy of 3 months and more
* given written informed consent

Exclusion Criteria:

* had previous exposure to pegfilgrastim or filgrastim
* had received systemic antibiotics within 72hrs of chemotherapy
* prior total cumulative lifetime exposure to doxorubicin more than 240 mg/m or epirubicin more than 600 mg/m

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2010-10; Primary Completion 2012-11 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Duration of grade 4 neutropenia(ANC<500mm3) for cycle 1 | in cycle 1
  Stage I: The difference in mean duration of grade 4 neutropenia between GCPGC 3.6mg and GCPGC 6mg is measured by check ANC in cycle I.
  Stage II : The difference in mean duration of grade 4 neutropenia between GCPGC which dose was determined at Stage I and Neulasta is measured by check ANC in cycle 1.

SECONDARY OUTCOMES:
Time to ANC recovery (≥2,000/mm3) after nadir in cycle 1 | in cycle 1
Depth of ANC nadir in cycle 1 | in cycle 1
Rates of Febrile neutropenia in all cycles | in all cycles
  Stage I: only in cycle 1; Stage II: in all cycles
Rates of severe neutropenia persisting more than 3 days in cycle 1 (only for Stage II) | in cycle 1
ANC values at Day 7 in all cycles (only for Stage II) | Day 7 in alll cycles
Rates of delay or dose-reduction of chemotherapy due to neutropenia (only for Stage II) | all cycles
Number of hospitalization due to febrile neutropenia in cycle 2 and after (only for Stage II) | in clycle 2-6
Number of intravenous antimicrobial treatments due to febrile neutropenia | in all cycles

OTHER OUTCOMES:
Incidence of antibody development in patients receiving GCPGC compared to Neulasta | 3 months after last treatment
Vital sign, Physical examination, Laboratory tests, Occurrence of adverse reactions | in all cycles

CONTACTS AND LOCATIONS:
Overall Officials: Do-Youn Oh, M.D., Ph.D., Principal Investigator — Seoul National University Hospital; Chang-Hee Lee, M.D., Ph.D., Study Director — Green Cross Corporation; Seock-Ah Im, M.D., Ph.D., Principal Investigator — Seoul National University Hospital
Locations (15):
- South Korea (15):
  - Chungbuk National University Hospital, Chungju, Chungchungbuk
  - National Cancer Center, Ilsan, KyungKi
  - Gachon University Gil Hospital, Incheon, KyungKi
  - Seoul National University Bundang Hospital, Sungnam, Kyungki
  - Keimyung University Dongsan medical Center, Daegu
  - Pusan National University Hospital, Pusan
  - Chung-Ang University Hospital, Seoul
  - Inha University Hospital, Seoul
  - Konkuk University Medical Center, Seoul
  - Kyung Hee University Medical Center, Seoul
  - Seoul Asan Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Seoul St.Mary's Hospital, Seoul
  - SMG-SNU Boramae Medical Center, Seoul
  - Ulsan University Hospital, Ulsan